CLINICAL TRIAL: NCT06822933
Title: The ReMonit Gout Study
Brief Title: The Remote Monitoring of Gout Study
Acronym: ReMonit Gout
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: Helse Sor-Ost (Other Government); The Dam Foundation (Other)
Responsible Party: Principal Investigator, Nina Osteras, Professor, Diakonhjemmet Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 861240; 24/04766 (Other: Diakonhjemmet Hospital)
Record Dates: First submitted 2025-02-07; First posted 2025-02-12 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Gout Initiating Urate-loweringUrate-lowering Therapy
Keywords: gout; randomised controlled trial; remote monitoring; eHealth; Urate-lowering Theraphy
MeSH Terms: conditions — Gout

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistical analyses will be conducted in line with the statistical analysis plan (SAP) by a biostatistician blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): State-of-the-art nurse-led treat-to-target follow-up strategy.
  Interventions: Other: Nurse-led follow-up with telephone consultations.
- Digital self-management (Experimental): Digital self-management strategy with patient self-management app, monthly blood tests, and remote monitoring by the study nurse until the treatment target is reached.
  Interventions: Device: Urika

INTERVENTIONS:
Device: Urika — Self-management application for patients with gout receiving urate lowering therapy. The 'Urika'-app includes films and written information about gout and gout management, reminders for blood-tests and medication, a visualisation of serum urate level over time, and an algorithm to calculate the medication drug-dose escalation. The app also includes a chat function and a secure web-platform for remote monitoring and communication between the participant and nurse. The study nurse will log into the web-platform on weekdays to check patient-reported side effects, adherence to medication, the current dose, and the need for a renewal of urate lowering therapy prescription.
  Arms: Digital self-management
Other: Nurse-led follow-up with telephone consultations. — Nurse-led follow-up in specialist healthcare with monthly blood tests and telephone consultations until the treatment target is reached.
  Arms: Usual care

SUMMARY:
The goal of this clinical trial is to: compare a new digital self-management treatment strategy to usual care, for patients with gout receiving urate lowering therapy in specialist healthcare. The digital self-management strategy consists of app-based remote follow-up with the 'Urica' app, and remote monitoring by a nurse. Usual care consists of state-of-the-art nurse-led treat-to-target follow-up, with regular telephone consultations. The main question the study aims to answer is:

Is the digital self-management strategy for patients with gout non-inferior compared to usual care in obtaining and maintaining a low serum urate level at 12 months.

DETAILED DESCRIPTION:
The trial is a non-inferiority, parallel-group, pragmatic, randomised controlled trial, with 24 months follow-up.

A 15% non-inferiority margin will be used.

Patients with gout will be recruited from the outpatient clinic at Diakohjemmet Hospital, Oslo, Norway. 168 adults with a gout diagnosis and serum urate level >360 μmol/L will be recruited and then randomised 1:1 to either usual care or digital self-management.

All participants will have a face-to-face consultation with a nurse prior to entering the study. The nurse will inform about gout and gout management strategy, the medication start-up dose, and the serum urate level treatment-target (<360 µmol/L, or <300 µmol/L for participants with tophi). All participants will take a monthly blood-test and increase their urate lowering medication dose until they reach the serum urate level treatment-target.

Usual care: Participants receiving usual care will have monthly telephone consultations with a nurse, who will inform about the medication dose for the next month.

Digital self-management: Participants receiving the digital self-management strategy will get help to download the 'Urika' -app, and instructions in how to use the app. They will register the following information in the app: the serum urate treatment target, type of urate lowering medication, side effects from medication, medical adherene, and the serum urate level from the monthly blood test. An algorithm in the app will calculate the medication drug-dose escalation. The study nurse will monitor the participants' progress through a secure web-platform.

All participants will answer digital questionnaires and take blood tests at baseline, 12 and 24 month follow-ups and answer a short digital questionnaire every 3 months.

A process end economic evaluation will be conducted alongside the trial. The process evaluation will include data from interviews with participants and nurses providing the interventions, and back-end data from the 'Urica'-app.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age at screening
* Patients with a clinical diagnosis of gout
* Patients who fulfil the ACR/EULAR classification criteria
* Serum urate level >360 µmol/L at inclusion
* At least 1 gout flare in the past 12 months
* Having a smartphone/tablet

Exclusion Criteria:

* Pregnant or breastfeeding
* Contraindication for urate lowering therapy
* Comedication azatioprin or 6-mercaptopurin
* Unstable medical conditions (e.g., uncontrollable hypertension, impaired liver function); known stage 3b or higher chronic kidney disease (estimated glomerular filtration (eGFR) rate/creatinine clearance <45 mL/min); severe infection or gastrointestinal bleed
* Major co-morbidities (e.g., malignancies, severe cardiovascular disease, severe diabetes mellitus, severe respiratory diseases)
* Psychiatric or mental disorders, alcohol abuse or other substance abuse, language barriers or other factors which makes adherence to the study protocol difficult

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with serum urate level below the treatment target | At 12 months after enrolment.
  The proportion with low serum urate level (<360/300 μmol/L) at 12 months. Serum urate level is collected from blood test results taken at the 12-month follow-up.

SECONDARY OUTCOMES:
Proportion of participants with serum urate level below the treatment target at 24 months | At 24 months after enrolment.
  The proportion with low serum urate level (<360/300 μmol/L) at 24 months. Serum urate level is collected from blood test results taken at 24-month follow-up.
Mean serum urate level | At 12 and 24 months after enrolment.
  The participants' mean serum urate level at 12 and 24 months. Serum urate level is collected from blood test results taken at 12 and 24 months follow-up.
Time to treatment target is reached | 1-24 months after enrolment.
  The mean time from enrolment to treatment target (serum urate level <360/300 μmol/L) is reached. Serum urate level is collected from blood test results conducted every month until the treatment target is reached. Analyses at 12 and 24 months.
Participant satisfaction with the follow-up care | At 12 months after enrolment.
  Participant satisfaction with the care, measured by one item from The Nordic Patient Experiences Questionnaire, with five point response options ranging from "Very satisfied" to "Very dissatisfied" at 12 months.

OTHER OUTCOMES:
Number of acute gout flares | From enrolment to end of study at 24 months.
  Number of participant-reported acute gout flares fulfilling the GAFFO criteria, i.e., fulfilment of at least 3 of 4 patient-reported criteria: patient-defined gout attack, pain at rest score of >3 on a 0-10 numeric rating scale, presence of at least one swollen joint, and presence of at least one warm joint. Self-reported every 3rd month in a digital questionnaire. Analyses at 12 and 24 months.
Side-effects of urate lowering therapy | From enrolment to 12 months.
  Number and type of participant-reported side-effects of urate lowering therapy. Self-reported every 3rd month in a digital questionnaire, during telephone consultations, or reported in the chat in the self-management app. Analyses at 12 months.
Adverse events | From enrolment to 12 months.
  Number and type of registered adverse events including serious adverse events, adverse device effects, and serious adverse device effects. Self-reported every 3rd month in a digital questionnaire, in telephone consultations, or reported in the chat in the self-management app. Analyses at 12 months.
Adherence to serum urate lowering therapy | From enrolment to end of study at 24 months.
  Participant-reported adherence to serum urate lowering therapy in the last week and the last month. The participants self-report the number of days they have missed taking their urate lowering medication in the last week and in the last month. Collected every 3rd month from enrolment to end of study at 24 months. Analyses at 12 and 24 months.
Medication adherence | At 12 and 24 months.
  Participant-reported adherence to medication using the Medication adherence report scale (MARS-5), which included 5 items with a 5-point Likert scale (1=always, 2=often, 3=sometimes, 4=rarely, 5=never) and score range 5-25. Score 25 is best outcome, and a score of 23-25 is considered adherent.
Knowledge of gout and recommended treatment | At Baseline, 12, and 24 months after enrolment.
  The Gout Knowledge Questionnaire, which includes 10 multiple choice questions assessing patients' knowledge on pathogenesis, treatment of acute gout attacks, and management of chronic gout. Score range: 0-10 (number of correct answers), score 10 is the best outcome
Beliefs about Medicines | At Baseline, 12, and 24 months.
  The Beliefs about Medicines Questionnaire (BMQ) - Specific. Comprises two 5-item subscales assessing beliefs about the necessity of prescribed medication (Specific-Necessity) and concerns about prescribed medication based on beliefs about the danger of dependence and long-term toxicity and the disruptive effects of medication (Specific-Concerns). Likert scale scored 1-5 per item. Scores for Specific-Necessity and for Specific-Concerns are calculated separately, and higher scores indicate stronger beliefs in the concepts of the sub-scale.
Health related quality of life | At Baseline, 12, and 24 months after enrolment.
  Health related quality of life measured by the EuroQol-5 Dimensions-5 Levels (EQ-5D-5L). The EQ-5D-5L is a generic and preference-weighted measure of health-related quality-of-life based on 5 dimensions: mobility, self-care, activities of daily life, pain, and anxiety/depression. For each dimension, the participant assesses 5 possible levels of problems (from no to severe, which is scored from 1 to 5, higher scores indicate worse outcome). EQ-5D index values will be calculated.
Overall health | At Baseline, 12, and 24 months after enrolment.
  Participant-reported general health is part of the EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) instrument, scored on a visual analog scale (VAS) 0-100, higher score indicates better general health.
Pain due to gout | At Baseline, 12, and 24 months.
  Pain in the past week due to gout self-reported on a 0-10 numeric rating scale. Higher scores indicate worse outcome.
Patient global assessment of disease activity | At Baseline, 12, and 24 months.
  Patient global assessment of disease activity self-reported on a 0-10 numeric rating scale. Higher scores indicate worse outcome.
Activity Impairment | At Baseline, 12, and 24 months.
  Work Productivity and Activity Impairment (WPAI), item no.6. Self-reported activity impairment, reported on a 0-10 numeric rating scale. Higher scores indicate worse outcome.
Estimated costs | From enrolment to end of study at 24 months.
  Estimated costs related to the interventions, healthcare utilisation and other associated costs, time off work and sickness absence. We will use participant-reported data on time off work and travel expenses, data from the intervention providers on time spent providing the interventions, and data from national registries on: healthcare consultations in primary and specialist health care, medication prescriptions, sickness absence, work assessment allowance, and disability benefits. Analyses at 12 and 24 months.
System usability | Experimental arm (digital self-management): At 12 months.
  System Usability Scale (SUS). Ten items scored on a 5-point Likert scale (Strongly disagree - Strongly agree, sum score 0-40, which is converted into 0-100, 100= best score). A SUS score above a 68 would be considered above average and anything below 68 is below average.
Satisfaction with the Urika app | Experimental arm (digital self-management): At 12 months.
  Satisfaction with the Urika app, includes one item rated on a 0-10 numeric rating scale ranging from "Very satisfied" to "Very dissatisfied".

CONTACTS AND LOCATIONS:
Overall Officials: Nina Østerås, Prof., Principal Investigator — Diakonhjemmet Hospital
Locations (1):
- Diakonhjemmet Hospital, Oslo, Please Select, Norway

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified IPD used in the results publications from the trial can be made available.
Time Frame: The IPD will be availabel from 2039
Access Criteria: The data will only be made available to researchers upon reasonable request. Data will only be provided after submission of a project plan outlining the reason for the request and the planned analyses. The request will have to be approved by the ReMonit Gout project group.